CLINICAL TRIAL: NCT04337723
Title: Implementation of Ankle Brachial Index Measurements and Wound, Ischemia, and Foot Infection Testing in Rural Health Clinics
Brief Title: Implementation of ABI and WIfI in Rural Health Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Misty Humphries, Associate Professor of Surgery, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1374497
Record Dates: First submitted 2020-04-01; First posted 2020-04-08 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Peripheral Arterial Disease; Diabetic Foot; Diabetes Mellitus
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Clinic participants will be taught how to do ABI testing and WIfI scoring to identify patients with PAD/DM disease for early vascular referral.
  Interventions: Behavioral: ABI/WIFI scoring

INTERVENTIONS:
Behavioral: ABI/WIFI scoring — The initial ABI training workshop will be coordinated by the non-physician clinic staff champion, and all non-provider clinic staff will be asked to participate. The PI and a research assistant will conduct a 1.5-hour telemedicine training session instructing clinical staff in ABI measurement and WIfI and scoring, using the clinical scoring sheet. Following didactic teaching, participants will perform ABI tests under the guidance of the PI/research assistant and with the support of other participants. During each part of the workshop, specific attention will be directed to pitfalls and technical errors of the test. A pre-post assessment will be used to ensure comprehension of key concepts and performance of the ABI and WIfI tools.

SUMMARY:
The objective of this project is to assess the fidelity and sustainability of in improving provider performance with Ankle Brachial Index (ABI) assessment and ulcer staging with the would ischemia foot infection (WIfI) tool for new patients with lower extremity ulcers due to peripheral artery disease (PAD) and diabetes mellitus (DM) at RHCs in the telemedicine network through a rural provider education program that is aligned with preexisting continuing medical education activities.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the educational program, an RHC must:

* already have telemedicine capabilities with the UC Davis CHT,
* be within 3 hours driving time form UC Davis Medical Center,
* have a lead practitioner willing to act as the clinic's point person for the proposed educational project, and
* have seen at least 10 patients in the prior 3 months with foot ulcers due to DM, PAD or combined disease.

Exclusion Criteria:

To be eligible for the project, a RHC must NOT:

* have a dedicated foot ulcer assessment program with on-site measurement of arterial perfusion, and
* be located within a 45 minute drive of a vascular surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
ABI/WIFI adoption | 6 months
  This outcome is a binary (yes/no) outcome of whether a clinic is performing ABI and WIfI testing 6 months after the original training and implementation assistance

SECONDARY OUTCOMES:
ABI/WIFI adaption and fidelity | 6 months
  This outcome is a qualitative outcome. The outcome is based on the use a modified Program Assessment Fidelity Tool developed by Cummins. This tool tracks programmatic and evaluative changes over time. The tool asks respondents to determine the What, How, To Whom, Where, and Who program changes occur with definitions for each category. The tool classifies changes by cause.
ABI/WIFI sustainability | 6 months
  To assess sustainability, we will collect the number of patients seen with lower extremity ulcers over a one-year period and the number of patients with ABI measurement performed. We will review charts for the number of patients with WIfI classification documentation at the clinical encounter.

CONTACTS AND LOCATIONS:
Overall Officials: Misty D Humphries, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided